CLINICAL TRIAL: NCT06701318
Title: Ultrasound Shear Wave Elastography for Assessing Muscle Stiffness in Parkinson's Disease Patients
Brief Title: Ultrasound Shear Wave Elastography in Parkinson's Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Romany Kamal Farah, Principal Investigator, Assiut University
Other Study IDs: Ultrasound SWE in Parkinson's
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease
Keywords: Ultrasound SWE; Parkinson disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson's patients group: Parkinson's disease diagnosed patients who meet the eligibility criteria and not complain of other neurological or musculoskeletal diseases that can affect muscle stiffness.
  Interventions: Device: Ultrasound shear wave elastography
- Healthy non Parkinson's group: Healthy age matched individuals who do not meet the criteria of Parkinson's disease diagnosis and not complain of other neurological or musculoskeletal diseases that can affect muscle stiffness.
  Interventions: Device: Ultrasound shear wave elastography

INTERVENTIONS:
Device: Ultrasound shear wave elastography — An ultrasound machine (GE LogiQ S8) equipped with SWE technology will be used. A high-frequency linear transducer will be used and The machine settings will be optimized for musculoskeletal applications.

SUMMARY:
Parkinson's disease (PD) is a progressive neurodegenerative disorder characterized by motor symptoms including muscle rigidity as one of major motor symptoms affecting quality of life of Parkinson's disease patients, thus we aim to assess and quantify muscle stiffness in those patients using Ultrasound shear wave elastography .

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive neurodegenerative disorder characterized by motor symptoms like tremors, bradykinesia, muscle rigidity, and postural instability, as well as various non-motor symptoms . While the exact cause of Parkinson's disease is not fully understood, it is thought to result from a combination of genetic and environmental factors, leading to the degeneration of dopamine-producing neurons in the brain . PD is the second most common neurodegenerative disorder after Alzheimer's disease, primarily affecting those over 60, with a higher prevalence in men . The disease significantly impacts quality of life due to progressive motor and non-motor disabilities, and while treatments can alleviate symptoms, there is currently no cure . Disease progression and prognosis vary, with advanced stages often leading to severe disability and reduced life expectancy .

Muscle rigidity, one of the major motor symptoms, refers to the increased resistance when muscles are passively stretched . Accurate assessment of muscle stiffness is essential for monitoring disease progression and evaluating therapeutic interventions .

Traditionally, clinical assessment tools like the Unified Parkinson's Disease Rating Scale (UPDRS), part III, are used to evaluate rigidity severity in PD patients . These assessments, involving manual joint movement and muscle palpation by professionals, are subjective and prone to error . Thus, there is a growing need for noninvasive, quantitative tools to assess muscle stiffness in PD patients .

Tools like electromyography (EMG) and myotonometry offer quantitative measurements . Ultrasound shear wave elastography (SWE) is another non-invasive technique that measures tissue stiffness by analyzing shear wave propagation. While SWE shows promise for various conditions, its application in PD-related muscle rigidity remains relatively unexplored .

ELIGIBILITY:
Inclusion Criteria:

* patient diagnosed with Parkinson's disease
* Age between 40-85 years
* No other neurological or musculoskeletal disorders affecting the examined limb muscles.

Exclusion Criteria:

* History of other neurological or musculoskeletal disorders affecting the examined limb muscles.
* History of significant trauma or surgery in the examined limb within the last year.
* patients with contraindications to ultrasound( such as open skin wounds or severe skin conditions in the area of interest).

Ages: 40 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any patients diagnosed with Parkinson's disease and meeting the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Quantification of muscle stiffness in the study groups. | Baseline
  The primary outcome will be the measurement of muscle stiffness using Ultrasound Shear Wave Elastography (SWE) and comparing muscle stiffness values between Parkinson's disease patients and healthy non Parkinson's controls.

SECONDARY OUTCOMES:
Correlation of the measured muscle stiffness with clinical severity of Parkinson's disease. | Baseline
  Secondary outcomes will include the correlation of muscle stiffness values with clinical severity scores, such as the Unified Parkinson's Disease Rating Scale (UPDRS). This will help to assess the relationship between increased muscle stiffness and the progression of Parkinson's Disease.

CONTACTS AND LOCATIONS:
Overall Officials: Afaf A. Hassan, Study Director — Professor; Radwa K. Abdel-Naser, Study Director — Assistant professor

REFERENCES:
- [Background] Khan AU, Akram M, Daniyal M, Zainab R. Awareness and current knowledge of Parkinson's disease: a neurodegenerative disorder. Int J Neurosci. 2019 Jan;129(1):55-93. doi: 10.1080/00207454.2018.1486837. Epub 2018 Nov 22. PMID 29883227
- [Background] Prajjwal P, Flores Sanga HS, Acharya K, Tango T, John J, Rodriguez RSC, Dheyaa Marsool Marsool M, Sulaimanov M, Ahmed A, Hussin OA. Parkinson's disease updates: Addressing the pathophysiology, risk factors, genetics, diagnosis, along with the medical and surgical treatment. Ann Med Surg (Lond). 2023 Aug 8;85(10):4887-4902. doi: 10.1097/MS9.0000000000001142. eCollection 2023 Oct. PMID 37811009
- [Background] Cui L, Hou NN, Wu HM, Zuo X, Lian YZ, Zhang CN, Wang ZF, Zhang X, Zhu JH. Prevalence of Alzheimer's Disease and Parkinson's Disease in China: An Updated Systematical Analysis. Front Aging Neurosci. 2020 Dec 21;12:603854. doi: 10.3389/fnagi.2020.603854. eCollection 2020. PMID 33424580
- [Background] Church FC. Treatment Options for Motor and Non-Motor Symptoms of Parkinson's Disease. Biomolecules. 2021 Apr 20;11(4):612. doi: 10.3390/biom11040612. PMID 33924103
- [Background] Bloem BR, Okun MS, Klein C. Parkinson's disease. Lancet. 2021 Jun 12;397(10291):2284-2303. doi: 10.1016/S0140-6736(21)00218-X. Epub 2021 Apr 10. PMID 33848468
- [Background] Yin L, Du L, Li Y, Xiao Y, Zhang S, Ma H, He W. Quantitative Evaluation of Gastrocnemius Medialis Stiffness During Passive Stretching Using Shear Wave Elastography in Patients with Parkinson's Disease: A Prospective Preliminary Study. Korean J Radiol. 2021 Nov;22(11):1841-1849. doi: 10.3348/kjr.2020.1338. Epub 2021 Aug 19. PMID 34431245
- [Background] Rovini E, Maremmani C, Cavallo F. How Wearable Sensors Can Support Parkinson's Disease Diagnosis and Treatment: A Systematic Review. Front Neurosci. 2017 Oct 6;11:555. doi: 10.3389/fnins.2017.00555. eCollection 2017. PMID 29056899
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] Kim MR, Yun JY, Jeon B, Lim YH, Kim KR, Yang HJ, Paek SH. Patients' reluctance to undergo deep brain stimulation for Parkinson's disease. Parkinsonism Relat Disord. 2016 Feb;23:91-4. doi: 10.1016/j.parkreldis.2015.11.010. Epub 2015 Nov 19. PMID 26686260
- [Background] Guerra A, D'Onofrio V, Ferreri F, Bologna M, Antonini A. Objective measurement versus clinician-based assessment for Parkinson's disease. Expert Rev Neurother. 2023 Jul-Dec;23(8):689-702. doi: 10.1080/14737175.2023.2229954. Epub 2023 Jul 6. PMID 37366316
- [Background] Drakonaki EE, Allen GM, Wilson DJ. Real-time ultrasound elastography of the normal Achilles tendon: reproducibility and pattern description. Clin Radiol. 2009 Dec;64(12):1196-202. doi: 10.1016/j.crad.2009.08.006. Epub 2009 Oct 8. PMID 19913130
- [Background] Kronlage C, Grimm A, Romano A, Stahl JH, Martin P, Winter N, Marquetand J. Muscle Ultrasound Shear Wave Elastography as a Non-Invasive Biomarker in Myotonia. Diagnostics (Basel). 2021 Jan 23;11(2):163. doi: 10.3390/diagnostics11020163. PMID 33498617